CLINICAL TRIAL: NCT00795067
Title: Relation of Circulating Endothelium-derived Microparticle to Carotid Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Hisashi Kai, Associate professor of Medicine, Kurume University
Other Study IDs: KurumeU-08060
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — platelet-poor plasma whole blood urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Carotid atherosclerosis group: Patients who undergo carotid ultrasound examination for carotid atherosclerosis screening

SUMMARY:
The investigators hypothesized that circulating endothelium-derived microparticle (EMP) may be a useful surrogate marker of atherosclerosis and future episode of cerebrovascular events. Peripheral blood is drawn at the time of carotid ultrasound examination. Circulating EMPs are counted using flow-cytometry. The correlation among circulating EMP, ultrasound findings, and atherosclerotic risk factors are determined by multiple stepwise regression analysis. The prevalence of cerebrovascular events is also determined during 3-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo carotid ultrasound examination for screening of atherosclerosis

Exclusion Criteria:

* Cerebrovascular events within the last 12 months
* Acute coronary syndrome, coronary and peripheral intervention within the last 6 months
* Uncontrolled heart failure
* Other severe systemic diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo carotid ultrasound examination for screening of atheroscrelosis
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The number of circulating EMPs | at the time of carotid ultrasound examination

SECONDARY OUTCOMES:
The occurrence of cerebrovascular and/or cardiovascular events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Imaizumi, MD, PhD, Study Chair — Kurume University
Locations (1):
- Kurume University Hospital, Kurume, Fukuoka, Japan